CLINICAL TRIAL: NCT02810626
Title: Application of Diffusion Tensor Imaging and Tractography in Pediatric Tumor Surgery
Brief Title: DTI & Tractography in Pediatric Tumor Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre (Other)
Collaborators: University of Western Ontario, Canada (Other); Synaptive Medical (Industry)
Responsible Party: Principal Investigator, Sandrine DeRibaupierre, Neurosurgeon, London Health Sciences Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UWO HSREB Ref#107499
Record Dates: First submitted 2016-03-18; First posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Brain Damage, Chronic; Cerebellar Cognitive Affective Syndrome; Cerebellar Mutism
MeSH Terms: conditions — Brain Damage, Chronic; Cerebellar Cognitive Affective Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Control Group (surgical standard of care): Subjects 18 years and younger diagnosed with a pediatric brain tumor, and who are eligible for surgical treatment will be recruited. All subjects will have clinical MRI scans that include a diffusion tensor imaging (DTI) protocol. Surgery will be carried out according to usual standard of care, without the use of processing for DTI tractography. Additional clinical scanning with the same protocol will be carried out post-operatively at 6 months. Pre-operative and post-operative quality of life assessments, functional testing and clinical outcome tests will be conducted at this post-operative period (6-months).
- Interventional (Other): Interventional Group (involvement of all BrightMatter™ products): Subjects 18 years and younger diagnosed with a pediatric brain tumor and who are eligible for surgical treatment will be recruited. All subjects will have clinical MRI scans that include a diffusion tensor imaging (DTI) protocol and will be sent to the interventional technology (BrightMatter Bridge) for quality control. The QC'ed images will then be sent to a pre-operating planning software (BrightMatter Plan) for planning the surgical approach. Surgery will be carried out with guidance from the exported plan and the intra-operative neuro-navigation software, BrightMatter Guide, with the use of post-processing DTI tractography. Additional clinical scanning with the same protocol will be carried out post-operatively at 6 months. Pre-operative and post-operative quality of life assessments, functional testing and clinical outcome tests will be conducted at this post-operative period (6-months).
  Interventions: Device: BrightMatter™ products

INTERVENTIONS:
Device: BrightMatter™ products — BrightMatter™ Plan (BMP): BMP is a software that enables surgeons to plan their neurosurgery preoperatively. BMP automatically generates whole brain tractography and highly accurate fusion of anatomical MRI and DTI images.
  BrightMatter™ Bridge (BMB):BMB involves offering SMI's MRI expertise to ensure a smooth workflow in neuroimaging including DTI to ensure optimized protocols are used to acquire the DTI images. Once the images are acquired, they are evaluated for their quality in real time using a quality control (QC) algorithm. The QC allows quality assessment of DTI images at the time-of-scan allowing for immediate correction while the patient is still there and reduces the need for patient re-scan.
  BrightMatter™ Guide (BMG): BMG is a neuro-navigation system that utilizes the DTI information and the trajectory planned by the surgeon in BMP pre-operatively, but bringing it into the operating room intraoperatively.
  Other Names: BrightMatter™ Plan, BrightMatter™ Bridge, BrightMatter™ Guide
  Arms: Interventional

SUMMARY:
The goal of this project will be to demonstrate that Synaptive Medical's Diffusion Tensor Imaging(DTI) product functionality used in pre-operative planning and intraoperative surgical navigation, improves clinical outcomes corresponding to a reduction in neurological and neuropsychological deficits in pediatric brain tumor surgery.

DETAILED DESCRIPTION:
Brain tumours are the most common form of solid tumours in children which often arise from the cerebellum. Treatment involves a complete resection of the tumour. Although surgical resection may eliminate most of the malignancy, signs of post-neurologic deficit may present as a consequence to the treatment.

One such example is cerebellar mutism syndrome (CMS), a postoperative syndrome typically arising 1 to 2 days after resection of a midline posterior fossa tumor; it consists of diminished speech progressing to mutism, emotional lability, hypotonia, and ataxia. While some of the symptoms recover after a few months, neuropsychological testing shows long term deficits in language (agramatism), executive function and verbal memory.

This study aims to investigate whether the use of Synaptive Medical's BrightMatter™ technology can help neurosurgeons better visualize and plan surgeries by avoiding eloquent fiber tracts in the brain and cerebellum; thus minimizing damage pertaining to neurologic and motor functionality. The use of these products will also be assessed for improved clinical outcomes in pediatric tumor surgery.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric subjects between the ages of 0-18 years with a brain tumor.

Exclusion Criteria:

* Pediatric subjects with contra-indication to MRI (metal, claustrophobia, etc.)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Total volume of tract damage | Assess the total volume of tract damage from baseline pre-operative examination through study completion (~ 1 year).
  Measure # of damaged tracts
Total size of craniotomy (resection zone) | Measure the total size of craniotomy from time of incision to end of surgery. (1 measurement/subject).
  Measure craniotomy size

SECONDARY OUTCOMES:
Total time it takes for the surgeon to pre-operatively plan cranial approach. | Assessed during start of surgical pre-operative plan through to end of surgical pre-operative plan (1 measurement/subject).
  Measured in hours
Total OR time | Assessed during surgical visit
  Measured in hours
Duration of hospital stay | Assessed during surgical visit up to 26 weeks
  Measured in # of days
Total cost of surgery | Assessed through study completion, an average of 1 year
Quality of life assessment | Assessed during surgical visit up to 26 weeks
  Measured using a standard questionnaire known as the WHOQOL-BREF questionnaire-World Health Organization Quality of Life Assessment
Functional testing | Assessed during surgical visit up to 26 weeks
  Measured using a routine functional impairment test for the pediatric population known as the Lansky performance scale
# deaths and complications with surgery | Assessed post-operatively after each surgery. Patient is followed until study completion (~ 1 year).
  Number of cases